CLINICAL TRIAL: NCT04105166
Title: Gene Therapy for Pyruvate Kinase Deficiency (PKD): A Phase I Clinical Trial to Evaluate the Safety of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the Codon Optimized Red Cell Pyruvate Kinase (coRPK) Gene in Adult and Pediatric Subjects With PKD
Brief Title: Gene Therapy for Pyruvate Kinase Deficiency (PKD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP-L301-0119
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pyruvate Kinase Deficiency
Keywords: hemolytic anemia; anemia; gene therapy
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic; Anemia

STUDY DESIGN:
Intervention Model Description: Initial safety evaluation will occur in an adult cohort (n=2) patients, followed by pediatric patients ages 8-17 (n=2-3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-L301 (Experimental): RP-L301 is a gene therapy product containing autologous genetically modified CD34+ hematopoietic stem cells containing the corrected PKD gene
  Interventions: Biological: RP-L301

INTERVENTIONS:
Biological: RP-L301 — Autologous genetically modified CD34+ hematopoietic stem cells containing the corrected PKD gene

SUMMARY:
This is an open-label Phase I trial to evaluate the safety of a hematopoietic cell-based gene therapy for patients with Pyruvate Kinase Deficiency (PKD).

DETAILED DESCRIPTION:
Autologous hematopoietic stem cells from mobilized peripheral blood will be transduced ex vivo (outside the body) with a lentiviral vector carrying a correct copy of the deficient PKD gene. The corrected stem cells will be infused intravenously back to the patient with the goal of correcting the hematological manifestations of the disease.

ELIGIBILITY:
Inclusion Criteria:

* PKD diagnosis with a confirmed PKLR mutation.
* Adult Cohort ≥18 years old and <50 years for the initial 2 patients enrolled; Pediatric Cohort ≥8-17 years for the next 2-3 patients.
* History of severe, transfusion-dependent anemia, defined as:

  1. At least 6 red blood cell transfusion episodes over a prior 12-month period and Hb levels <9.5 g/dL in the previous 12 months despite splenectomy OR
  2. At least 3 red blood cell transfusion episodes per year over 2 prior years (in the absence of precipitating events such as infection or surgery) and Hb levels <9.5 g/dL in the previous 12 months despite prior splenectomy.

     OR
  3. Hb levels <8.0 g/dL despite prior splenectomy in the absence of transfusions (documented during 2 or more assessments during the prior 1-2 years) regardless of transfusion requirements.
* Adequate cardiac, pulmonary, renal and hepatic function, as detailed in relevant exclusion criteria.
* Availability of detailed medical records, including transfusion requirements, for at least the prior 2 years.
* Willing and able to read and correctly understand the patient information sheet and provide consent (or informed assent for minors) regarding study participation.
* Negative serum pregnancy test for female patients of childbearing potential.

Exclusion Criteria:

* Presence of other known causes of hemolysis (in addition to PKD). Patients with concurrent G6PD deficiency diagnosed during pre-study evaluation may be considered for eligibility if in the opinion of the Investigator, the hemolytic anemia is the result of PKD and the G6PD deficiency is considered an incidental finding.
* A venous thromboembolic event (VTE; i.e., pulmonary embolism or deep vein thrombosis) or arteriothromboembolic event (ATE; including unstable angina, myocardial infarction, stroke or transient ischemic attack) during the prior 12 months.
* Any evidence of severe iron overload that, per Investigator discretion, warrants exclusion.
* Evidence of bridging fibrosis, cirrhosis or active hepatitis on liver biopsy. Liver biopsy is required when liver iron concentration (LIC) is ≥15 mg/g on T2* magnetic resonance imaging (MRI) of liver. If a liver biopsy has been performed less than 6 months prior to enrollment, it does not need to be repeated.
* Significant medical conditions including documented HIV infection, active viral hepatitis, poorly-controlled hypertension, pulmonary hypertension cardiac arrhythmia or congestive heart failure; pulmonary hypertension or ATEs (including stroke or myocardial infarction) within the 6 prior months.
* Active hematologic or solid organ malignancy, not including non-melanoma skin cancer or another carcinoma in situ. Patients with previously resected solid organ malignancies or definitively treated hematologic malignancies may be eligible if there has been no evidence of active malignancy during the prior 3 years.
* Uncontrolled seizure disorder.
* Cardiac T2*<10 ms by magnetic resonance imaging (MRI) or left ventricular ejection fraction (LVEF) <45% by echocardiogram or multiple gated acquisition (MUGA) scanning.
* Hepatic dysfunction as defined by: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5× the upper limit of normal.(ULN).
* Renal dysfunction as defined as serum creatinine > ULN. Patients with creatinine above ULN may be eligible pending documentation of a GFR ≥60 mL/min/1.73m2 as calculated by the Modification of Diet in Renal Disease equation (Stevens 2006), the revised Schwartz formula (for patients under 18 years old) (Schwartz 2009), or 24-hour urine collection.
* Pulmonary dysfunction as defined by either:

  * Need for supplemental oxygen during the prior 2 weeks (in absence of acute infection) or
  * Oxygen saturation (by pulse oximetry) <90%.
* Any medical or other contraindication for both leukapheresis and BM harvest procedure as determined by the treating Investigator.
* Any medical or psychiatric condition that in the opinion of the Investigator renders the subject unfit for trial participation or at higher than acceptable risk for participation.
* Poor functional status, evidenced by Karnofsky Index <70 in adults or Lansky <70 in children.
* Participation in another clinical trial with an investigational drug within 14 days before the informed consent signature. Participation in observational studies is allowed.
* Pregnant women or women with a positive serum pregnancy test at screening or breast feeding or planning to become pregnant within the next 24 months. Women not willing to use highly effective contraceptive methods during the complete study period.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and toxicity of RP-L301: number of participants with treatment-related adverse events | 2 years
  The number of participants with treatment-related adverse events as assessed by United States (US) National Cancer Institute (NCI) v.5.0.

SECONDARY OUTCOMES:
Genetic correction following administration of RP-L301 | 2 years
  Evidence of multi-lineage gene correction in peripheral blood (PB) and bone marrow (BM cells) will be assessed by measuring vector copy number
Transfusion independence | 1 year
  Transfusion independence (when relevant) at 12 months defined as need for less than or equal to 1 red blood cell transfusion in the previous 6 months
Reduction in transfusion requirements | 1 year
  50% reduction in transfusion requirements (when relevant) at 12 months (assessed in the previous 6 months for the 12-month assessment) relative to the 1-year period prior to enrollment
Clinically significant reduction in anemia | 2 years
  Increase in pre-transfusion hemoglobin (Hb) levels of 1.5 g/dL (determined by 2 assessments separated at least three months over the first and second year of follow up) relative to the average of patient's Hb levels before blood transfusions over the year prior to enrollment OR
  Increase of at least two-fold in the time to pre-transfusion Hb nadir relative to the average transfusion interval over the year prior to enrollment, where pre-transfusion Hb nadir is defined as the average Hb value (during the year prior to enrollment) prior to red blood cell (RBC) transfusions
Reduction of hemolysis | 1 year
  Reduction of reticulocytosis, defined as the number of patients with a reduction of 50% from the average of a patient's absolute reticulocyte counts (obtained prior to therapeutic blood transfusions) over the year prior to enrollment at 12 months subsequent to investigational therapy

CONTACTS AND LOCATIONS:
Overall Officials: José Luis López Lorenzo, MD, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz; Ami Shah, MD, Principal Investigator — Stanford University; Julián Sevilla Navarro, MD, PhD, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz
Locations (3):
- Stanford University, Stanford, California, United States
- Spain (2):
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: Undecided